CLINICAL TRIAL: NCT07156721
Title: The Effect of Using a White Reflective Drape During Phototherapy on Bilirubin Levels and Hospital Stay in Neonates
Brief Title: White Reflective Drape in Phototherapy for Neonatal Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sıla İpek DURMUŞ, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaglikBilimleriU-SID-01; 2023/122 (Other: Gülhane Clinical Research Ethics Committee)
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Phototherapy; White Reflective Drape; Bilirubin; Jaundice; Newborn; Neonatal Intensive Care; nursing
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: This was a randomized controlled trial with two parallel groups. Participants were randomly assigned to either the intervention group (phototherapy with a white reflective drape) or the control group (standard phototherapy). Groups were treated simultaneously and outcomes compared at baseline, 4 hours, and 24 hours.
Masking Description: This was an open-label study; no masking was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - White Reflective Drape (Experimental): Neonates received phototherapy with a white reflective drape placed around three sides and overhead of the device, and a white sheet placed under the infant to increase light reflection.
  Interventions: Device: Phototherapy with White Reflective Drape
- Control Group - Standard Phototherapy (Active Comparator): Neonates received standard phototherapy without a white reflective drape or additional reflective materials.
  Interventions: Device: Standard Phototherapy

INTERVENTIONS:
Device: Phototherapy with White Reflective Drape — Phototherapy device (24 blue LED, 1 red LED, Ertunç Özcan) at 35 cm distance; a double-layer white reflective drape (125 × 105 cm) was placed around three sides and overhead, with a white sheet under the infant.
  Arms: Intervention Group - White Reflective Drape
Device: Standard Phototherapy — Phototherapy device (24 blue LED, 1 red LED, Ertunç Özcan) at 35 cm distance; no reflective drape or additional reflective material used.
  Arms: Control Group - Standard Phototherapy

SUMMARY:
This randomized controlled trial investigated the effect of using a white reflective drape during phototherapy on serum bilirubin levels and hospital stay in neonates diagnosed with hyperbilirubinemia. A total of 102 newborns (≥34 weeks gestational age) were randomized into two groups: an intervention group (phototherapy with a white reflective drape) and a control group (standard phototherapy). Serum bilirubin levels were measured at baseline, 4 hours, and 24 hours. The primary outcome was the reduction in serum bilirubin at 24 hours, and secondary outcomes included bilirubin reduction rates at different time intervals, phototherapy duration, and hospital stay.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia is one of the most common conditions in the neonatal period and may lead to severe complications if untreated. Phototherapy is the standard treatment; however, its effectiveness can be improved by using reflective materials to enhance light exposure.

In this single-center randomized controlled trial, conducted between October 2023 and August 2024 at the Neonatal Intensive Care Unit of a University Hospital in Ankara, Turkey, a total of 102 neonates with hyperbilirubinemia were enrolled. Inclusion criteria were: gestational age ≥34 weeks, diagnosis of hyperbilirubinemia, physician decision to initiate phototherapy, and written parental consent. Exclusion criteria included critical health conditions (e.g., Extracorporeal membrane oxygenation or nitric oxide therapy), congenital anomalies, blood group incompatibility or positive Coombs test, and bilirubin at exchange transfusion threshold.

Participants were randomized into two groups (n=51 per group). In the intervention group, a white reflective drape made of double-layer alpaca fabric (125 × 105 cm) was placed around the phototherapy device (three sides plus overhead) and a white sheet was placed under the neonate. The control group received standard phototherapy without a reflective drape. Phototherapy was administered using an Ertunç Özcan device with 24 blue LED lamps and one red focusing light. Serum bilirubin levels were measured from capillary blood samples at baseline, 4 hours, and 24 hours, maintaining a device-to-infant distance of 35 cm.

The primary outcome was the change in serum bilirubin at 24 hours. Secondary outcomes included bilirubin reduction rates (0-4h, 4-24h, 0-24h), phototherapy duration, and hospital length of stay. Statistical analysis was performed using SPSS v23, applying t-test, Mann-Whitney U, Friedman, and Dunn's tests, with significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 34 weeks
* Diagnosed with hyperbilirubinemia
* Physician decision to initiate phototherapy Written informed consent obtained from parents

Exclusion Criteria:

* Critical illness (e.g., ECMO, nitric oxide therapy)
* Congenital anomalies
* Blood group incompatibility or positive Coombs test
* Bilirubin level at exchange transfusion threshold

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Change in serum bilirubin level at 24 hours | 24 hours
  Serum bilirubin level measured at baseline and at 24 hours after initiation of phototherapy.

SECONDARY OUTCOMES:
Change in serum bilirubin level at 4 hours | 4 hours
  Serum bilirubin level measured at baseline and at 4 hours.
Bilirubin change rate between 0-4 hours | 0-4 hours
  Percentage change in bilirubin from baseline to 4 hours.
Bilirubin change rate between 4-24 hours | 4-24 hours
  Percentage change in bilirubin from 4 to 24 hours.
Bilirubin change rate between 0-24 hours | 0-24 hours
  Percentage change in bilirubin from baseline to 24 hours.
Duration of phototherapy | Up to 72 hours
  Total duration of phototherapy administered until bilirubin decreased below treatment threshold.
Hospital length of stay due to hyperbilirubinemia | Up to 7 days
  Total hospitalization duration (hours) from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Berna EREN FİDANCI, Assoc. Prof. Dr., Principal Investigator — Gülhane Faculty of Nursing, Child Health and Disease Nursing Department
Locations (1):
- Gazi University Hospital, Neonatal Intensive Care Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No